CLINICAL TRIAL: NCT07298967
Title: ORegon CHild Absenteeism Due to Respiratory Disease Study - Air Surveillance
Brief Title: ORCHARDS-AIR Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2025-1617; AS (Other: UW Madison); UWMSN | SMPH | DFMCH Departmen (Other: UW Madison); Protocol Version 12/15/2025 (Other: UW Madison)
Record Dates: First submitted 2025-12-19; First posted 2025-12-23 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-12

CONDITIONS: Acute Respiratory Infection; Influenza-like Illness

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Students with ARI (acute respiratoy infection) (Experimental): Students with ARI and their household members will provide nasal swabs
  Interventions: Diagnostic Test: Nasal swab; Device: Indoor air quality monitor

INTERVENTIONS:
Diagnostic Test: Nasal swab — Participants will use a swab to collect nasal specimens
Device: Indoor air quality monitor — InBio Apollo ambient air sampler to be run in the home for the duration of study participation. Material from the air, like aerosols, dust particles, and other environmental material, are collected on sampler filler material.

SUMMARY:
The purpose of this observational study is to compare the effectiveness of air surveillance and to better understand the relationship between household transmission and viruses detected in the air.

Participants will provide nasal swabs and have an air sample surveillance device installed in their home.

DETAILED DESCRIPTION:
The purpose of ORCHARDS-AIR is to utilize air surveillance in participant homes in conjunction with individually collected nasal specimens to assess their concordance and evaluate the significance of airborne detection with household transmission of common respiratory pathogens such as influenza and SARS-CoV-2.

The researchers postulate that households with documented and probable respiratory pathogen transmission will have higher rates of in-home air surveillance detection. Students with more severe illnesses will be absent more often and spend more time at home, potentially leading to absenteeism being associated with greater air surveillance detections and intrahousehold transmission.

ELIGIBILITY:
Inclusion Criteria - Students:

* Student attends, or is eligible to attend, a school within the Oregon School District (OSD)
* Study has an illness characterized by at least 2 of 6 acute respiratory infection (ARI)/ILI symptoms (nasal discharge, nasal congestion, sneezing, sore throat, cough, fever) and student scores at least 2 points on the Jackson scale

Exclusion Criteria - Students:

* Household member listed on Wisconsin Department of Corrections Sex Offender Registry
* Illness onset more than 7 days before anticipated time of specimen collection
* Anatomical defect for which nasal specimen collection is contraindicated
* Student participated too recently (<7 days from day 14 during peak influenza / COVID-19 period and <30 days during other times, as determined by a medically-attended surveillance program)

Inclusion Criteria - Household member:

* Live in the same household as eligible student participant
* Any age and gender
* Fluent in English
* Able to provide appropriate consent or assent

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 422 (Estimated)
Dates: Start 2026-01-07 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Rate of virus detection | Day 0, Day 7, Day 14
  Participants will provide nasal swabs, which will be tested for a panel of viruses.
Rate of air sampling detection among families with documented transmission | Day 7, Day 14
  Study team will collect and test air sampler filter for viruses.
Rate of air sampling detection among families without documented transmission | Day 7, Day 14
  Study team will collect and test air sampler filter for viruses.
Survey of symptoms - day 0 | Day 0
  Qualitative survey of participants' symptoms and related activities.
Survey of symptoms - day 7 | Day 7
  Qualitative survey of participants' symptoms and related activities.
Survey of symptoms - day 14 | Day 14
  Qualitative survey of participants' symptoms and related activities.
Air sampler use survey | Day 7, Day 14
  Qualitative survey about participants' use of the air sampler.

SECONDARY OUTCOMES:
Number of absences | 14 days
  Participants will self-report whether they were absent from school during the study period.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Temte, MD, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin-Madison, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes